CLINICAL TRIAL: NCT06068205
Title: COMPARATIVE ANALYSIS OF THE MORPHO-MECHANICAL PROPERTIES OF RED BLOOD CELLS EXTRACTED FROM DIABETIC PATIENTS WITH AND WITHOUT MICROVASCULAR COMPLICATIONS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5860
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetes with microvascular complications
  Interventions: Diagnostic Test: Blood test - atomic force microscopy in the force spectroscopy mode
- Type 1 diabetes without microvascular complications
  Interventions: Diagnostic Test: Blood test - atomic force microscopy in the force spectroscopy mode

INTERVENTIONS:
Diagnostic Test: Blood test - atomic force microscopy in the force spectroscopy mode — A single blood test to be analysed through atomic force microscopy in the force spectroscopy mode

SUMMARY:
The aim of the study is to analyse the biomechanical stiffness of red blood cells extracted from subjects with type I diabetes with and without microvascular complications through a biophysical characterization of red blood cells using microscopy, spectroscopy and scattering measurements. 48 subjects with type 1 diabetes, 24 with and 24 without microvascular complications will be enrolled. From all subjects a single blood sample will be taken to perform the analysis of red blood cells morpho-mechanical properties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes for at least 10 years
* Stable metabolic control (HbA1c <7.5%) for at least 6 months
* BMI between 18.5 and 30 Kg/m^2
* Systolic blood pressure < 140 mmHg and diastolic blood pressure <90 mmHg

Exclusion Criteria:

* Blood pressure higher than 140/90 mmHg
* Unstable metabolic control (HbA1c >7.5%)
* BMI > 30 Kg/m^2 or < 18.5 Kg/m^2
* Liver failure
* Concomitant acute infections
* Uncontrolled thyroid diseases
* Pregnancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type I diabetes mellitus with (case group) and without (control group) microvascular complications. The two groups will be balanced for age (50-70 years), age of disease (>10 years), glycaemic control and BMI value.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-09-29 (Estimated); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
In 48 subjects with type 1 diabetes with and without microvascular complications, the average stiffness of red blood cells, measured using atomic force microscope and quantified using Young's modulus, will be measured. | 1 day
  Young's modulus values are obtained using atomic force microscopy